CLINICAL TRIAL: NCT01172717
Title: Phase II Study of Panitumumab in the Treatment of Carcinoid Syndrome
Brief Title: Study of Panitumumab in the Treatment of Carcinoid Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never began
Sponsor: Boston Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31701
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Carcinoid Syndrome
Keywords: Carcinoid; Carcinoid syndrome
MeSH Terms: conditions — Serotonin Syndrome; Carcinoid Tumor | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab (Experimental): Single arm study
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Panitumumab will be given by intravenous infusion at a dose of 9 mg/kg on day 1 of study and then every 3 weeks until progression of disease
  Other Names: Vectibix; ABX-EGF

SUMMARY:
The primary hypothesis of this study is that panitumumab, an inhibitor of the epidermal growth factor receptor (EGFR), is an effective treatment for carcinoid syndrome in people who fail or do not adequately respond to octreotide or other supportive therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic carcinoid tumor and carcinoid syndrome
* Measurable disease as defined by RECIST criteria or evaluable disease

  1. Measurable disease is the presence of at least one measurable lesion. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions are lesions that can be accurately measured in at least one dimension with longest diameter greater than or equal to 20 mm using conventional techniques or greater than or equal to 10 mm with spiral CT scan.
  2. Evaluable disease is disease that cannot be measured directly by the size of the tumor but can be evaluated by a validated biomarker assay including 24 hr urine 5-hydroxyindoleacetic acid, serum serotonin, and/or serum chromogranin A.
  3. All sites of disease must be evaluated less than or equal to 28 days prior to enrollment.
* All subjects must be 18 years of age or older.
* ECOG performance status of 0 to 2.
* Subjects may have had past or may be receiving current treatment with octreotide.
* Adequate laboratory parameters with all tests to be performed within 72 hours prior to the first dose.

  1. Absolute neutrophil count greater than or equal to 1.5 x 109/L
  2. Hemoglobin greater than or equal to 9.0 g/dL
  3. Platelet count greater than or equal to 100 x 109/L
  4. Serum creatinine less than 1.5 mg/dL
  5. Aspartate aminotransferase (AST) less than or equal to 3 times the upper limit of normal, unless with radiographic evidence of liver metastases. If with liver metastases, AST less than 5 times the upper limit of normal.
  6. Alanine aminotransferase (ALT) less than or equal to 3 times the upper limit of normal, unless with radiographic evidence of liver metastases. If with liver metastases, AST less than 5 times the upper limit of normal.
  7. Total Bilirubin less than or equal to 1.5 times the upper limit of normal.
  8. Magnesium level greater than lower limit of normal
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Woman and men should use adequate birth control for at least 6 months after the last administration of panitumumab.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Evidence of localized carcinoid tumor amenable to surgical resection or chemoembolization.
* People who are asymptomatic from their carcinoid tumors.
* Past treatment with EGFR inhibitors including cetuximab and panitumumab.
* History of active malignancies requiring treatment in the past 5 years with the exception of resected basal cell carcinoma of the skin.
* History of interstitial pneumonitis or pulmonary fibrosis.
* History of cardiac arrhythmia or Q-T prolongation on electrocardiogram.
* Women who are pregnant or breast feeding.
* Known infection with human immunodeficiency virus (HIV).
* Treatment with chemotherapy, biologics, immunotherapy, vaccines or cytokine therapy within 4 weeks prior to study entry. The use of octreotide is not exclusionary.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of enrollment.
* A negative octreotide scan does not exclude study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Radiographic measures | Every 4 cycles
Tumor Marker Evaluations | Every 2 cycles

SECONDARY OUTCOMES:
Quality of LIfe | Day 1 each cycle and 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kevan Hartshorn, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts